CLINICAL TRIAL: NCT00526539
Title: Is There Increased Polyethylene Wear and Increased Periprosthetic Bone Loss in Femur in Reverse Hybrid Technique Compared With Conventional Cemented Technique in Total Hip Replacement?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Reverse hybrid vs cemented THR
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2007-09

CONDITIONS: Osteoarthritis
Keywords: THR; reversed hybrid; wear
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement, Hip

INTERVENTIONS:
Other: Total hip replacement, Spectron and Taperloc

SUMMARY:
Total hip replacement is a very cost effective procedure to enhance life quality in a group of patients. In the period 2000-2004 7-8000 procedures were preformed, 13% were revisions (1). Historically, many different principles have been used from the first resurfacings to cemented and uncemented total hip replacements as we know them today. In 2000, 28 different femoral stems and 26 different acetabular components were in regular use in Norway. There are several well-documented cemented acetabular components, but no such uncemented cup. On the femoral side there are several well-documented stems both cemented and uncemented. (2).

From the late 1990's a reverse hybrid (uncemented stem and cemented cup) is being more frequently used. In 2004 a total of 276 reverse hybrid hips were done and the trend is increasing. (1). This technique is solely based on experience and the fact that one combines the better of two principles (cemented and uncemented). There is no scientific evidence that this technique is as good or better than a cemented THR.

One of the potential problems with hydroxyapatite coated components is that it is suspected that it may increase wear due to the particle theory. (3,4). There are no prospective randomised controlled RSA and DXA studies that conclude on this matter. This is such a study and our hypothesis is that there is no difference in wear or osteolysis between the methods.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis
* Indication for THR

Exclusion Criteria:

* Significant anatomical abnormalities
* Rheumatoid artheritis, dysplasia, fracture sequela

Max Age: 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Lars Nordsletten, professor, MD, Ph.D, Study Chair — Ullevål University Hospital, N-0407 Oslo; Einar Lindalen, MD, Principal Investigator — Lovisenberg Hospital, N- 0440 Oslo